CLINICAL TRIAL: NCT05511649
Title: The Prognostic Impacts and Clinical Utility of the Characteristics of New-onset Atrial Fibrillation Complicating Acute Myocardial Infarction in China
Brief Title: New-Onset Atrial Fibrillation Complicating Acute Myocardial Infarction in China
Acronym: NOAFCAMI-China
Status: Completed | Type: Observational
Sponsor: Shanghai 10th People's Hospital (Other)
Collaborators: Kaifeng Central Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, Chief Physician, Shanghai 10th People's Hospital
Other Study IDs: NOAFCAMI-China
Record Dates: First submitted 2022-08-20; First posted 2022-08-23 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: New Onset Atrial Fibrillation; Acute Myocardial Infarction
Keywords: myocardial infarction; new-onset atrial fibrillation; atrial fibrillation burden; mortality
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post-MI NOAF with low AF burden: Patients with post-MI NOAF who had a AF burden<10.87%. The cut-off value of AF burden of 10.87% was identified based on our previous work.
  Interventions: Device: continuous electronic monitor
- Post-MI NOAF with high AF burden: Patients with post-MI NOAF who had a AF burden≥10.87%.
  Interventions: Device: continuous electronic monitor

INTERVENTIONS:
Device: continuous electronic monitor — All patients with MI hospitalized in the CCU department of Shanghai Tenth People's Hospital, KaiFeng Central Hospital, and the First Affiliated Hospital of Zhengzhou University will receive 24-hour continuous cardiac monitoring until discharge.
  Other Names: Philips IntelliVue MP40, Netherlands

SUMMARY:
To investigate the prognostic impacts of the atrial fibrillation burden (AFb) in acute myocardial infarction (AMI) patients who developed paroxysmal new-onset atrial fibrillation (NOAF) during the index AMI hospitalization.

DETAILED DESCRIPTION:
In the present study, investigators retrospectively reviewed the medical records of all acute MI patients who were admitted to the coronary artery unit (CCU) of Shanghai Tenth People's Hospital, KaiFeng Central Hospital, and the First Affiliated Hospital of Zhengzhou University between January 2014 and January 2022. All patients will routinely receive continuous electronic monitoring (CEM) throughout their hospital stay to detect cardiac arrhythmias including the AF events. Of these, patients with AMI without a history of AF who developed a first documented AF episode will be considered for inclusion. The AFb is measured as a percentage (%) by dividing the total AF duration by the total CEM duration.

ELIGIBILITY:
Inclusion Criteria:

1. Patients hospitalized for AMI including both STEMI and NSTEMI between January 2014 and January 2022 at the CCU department of Shanghai Tenth People's Hospital, KaiFeng Central Hospital, and the First Affiliated Hospital of Zhengzhou University.
2. Patients who developed a first documented AF (NOAF) during the index AMI hospitalization；
3. Adult patients (>18 years old).

Exclusion Criteria:

1. Patients with a medical history of pre-existing AF;
2. Patients with a medical history of rheumatic valvular disease;
3. Patients with a medical history of sick sinus syndrome;
4. Patients undergoing emergent coronary artery bypass surgery;
5. Patients' medical records with serious deficiencies and CEM data cannot be retrieved;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with post-MI NOAF
Sampling Method: Probability Sample
Enrollment: 832 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-09-23 (Actual)

PRIMARY OUTCOMES:
All-cause death | From the time of AMI discharge until occurrence of an outcome of interest, death, or loss to follow up, maximum up to 10 years
  Death from any cause

SECONDARY OUTCOMES:
Cardiovascular death | From the time of AMI discharge until occurrence of an outcome of interest, death, or loss to follow up, maximum up to 10 years
  Death from cardiovascular causes
Recurrent myocardial infarction | From the time of AMI discharge until occurrence of an outcome of interest, death, or loss to follow up, maximum up to 10 years
  Rehospitalization for myocardial infarction
Heart failure hospitalization | From the time of AMI discharge until occurrence of an outcome of interest, death, or loss to follow up, maximum up to 10 years
  HF hospitalization was based on clinical symptoms such as dyspnea and fatigue, and signs of peripheral or pulmonary edema that required hospitalization for intravenous diuretic treatment
Ischemic stroke | From the time of AMI discharge until occurrence of an outcome of interest, death, or loss to follow up, maximum up to 10 years
  Ischemic stroke was identified as the presence of a new focal neurologic deficit thought to be ischemic in origin, with signs or symptoms lasting> 24 hours, and was validated according to radiographic imaging test.
Major bleeding | From the time of AMI discharge until occurrence of an outcome of interest, death, or loss to follow up, maximum up to 10 years
  Bleeding event with a Bleeding Academic Research Consortium (BARC) classification of types 3 or 5.

CONTACTS AND LOCATIONS:
Overall Officials: Yidong Wei, M.D., Ph.D., Principal Investigator — Shanghai 10th People's Hospital
Locations (3):
- China (3):
  - KaiFeng Central Hospital, Kaifeng, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Luo J, Qin X, Yuan Y, Zhang Y, Liu J, Wang Y, Zhao G, Xiao L, Zhang X, Fang Y, Shi W, Qin L, Liu B, Wei Y; NOAFCAMI-China Registry Investigators. Association of Atrial Fibrillation Burden With Cardiovascular Outcomes in New-Onset Atrial Fibrillation Complicating Myocardial Infarction. J Am Heart Assoc. 2025 May 20;14(10):e039547. doi: 10.1161/JAHA.124.039547. Epub 2025 Apr 16. PMID 40240944